

## **INFORMED CONSENT FORM**

## **CAROPROT** – INFLUENCE OF PROTEINS ON CAROTENOID BIOAVAILABILITY

| | _, nereby acknowledge that I was informed in detail |
|---|---|
| about the present study. I was given enough infor | mation about its contents, objectives and about my |
| rights as a participant. | |
| I understood the information that was give | n to me; I had the opportunity to pose questions, |
| which were answered to my satisfaction. | |
| | samples in the study and I agree with the collection: |
| <ul><li>of blood and urine samples,</li></ul> | |
| □ of stool samples, | |
| | and analysis of samples is foreseen, as well as the |
| intake of additional proteins. The purpose and pos | |
| I am aware that some blood analyses will ha<br>the Clinical and Epidemiological Investigation Cent | ve to be carried out in other institutions outside of |
| | ill be treated in a strictly confidential way and it will |
| - , , | s, as written in the amended law of 2 <sup>nd</sup> August 2002 |
| on personal data protection. | , as written in the amenaca law of 2 Magast 2002 |
| · | of the results, in scientific journals, in complete |
| anonymity. | or the results, in scientific journals, in complete |
| | cipation from this study at any time after notifying |
| the project director, without compromising any fu | |
| | Consent Form. I sign it freely and voluntarily, and I |
| was given a signed copy of this document. | consent rorm. r sign it freely and voluntarily, and r |
| was given a signed copy of this document. | |
| Signature of Participant: | Date: |
| Part for the researcher: | |
| I hereby certify, | , having informed the |
| above participant about the objectives, the nature | e, the duration and the risks of this study and certify |
| that he / she agreed to take part in this study. | |
| Date: | Signature: |
| CONTACTS FOR FUR | THER INFORMATION |
| Jean-Yves Ferrand | Dr. Torsten BOHN |

Jean-Yves Ferrand (CIEC-LIH)

1A, rue Thomas Edison L-1445 Strassen Tel.: (+352) 26 970 800

e-mail: <u>jean-yves.ferrand@lih.lu</u>

(EPHRU-LIH)
1 A, rue Thomas Edison

L-1445 Strassen
Tel.:(+352) 26 970 394

e-mail: torsten.bohn@lih.lu